CLINICAL TRIAL: NCT06318624
Title: Immediate Effects of Ankle Mobilization With Movement and Mulligan Talocrural Taping on Gait and Balance in Stroke Patients
Brief Title: Immediate Effects of Ankle MWM and Taping on Gait and Balance in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Ismail Okur, Asst. Prof., Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KHSU-2023/11
Record Dates: First submitted 2024-02-14; First posted 2024-03-19 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Stroke
Keywords: stroke; gait; mobilisation; Mulligan; balance
MeSH Terms: conditions — Stroke | interventions — Movement; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Masking Description: There are 2 different groups in the study. One of them is the intervention group and the other is the sham group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Movement with Motion technique of Mulligan Concept to the ankle joint and taping will be performed on the participants in the Intervention Group.
  Interventions: Other: Mobilisation with Movement and Taping
- Sham Group (Sham Comparator): Movement with Motion technique of Mulligan Concept to the ankle joint with lower amplitude and taping with minimal tension will be performed on the participants in the Sham Group.
  Interventions: Other: Sham

INTERVENTIONS:
Other: Mobilisation with Movement and Taping — For MWM for the talocrural joint, the hemiparetic side of the participant is positioned in a standing position on a stool. A non-elastic belt is passed behind the patient's distal tibia and secured around the therapist's pelvis. The patient is asked to perform active knee flexion and ankle dorsiflexion with weight on the hemiparetic side. Meanwhile, the therapist performs forward sliding of the tibia with the help of the belt. For 10 seconds active and painless sliding takes place and then return to the starting position. This application is applied as 10 repetitions, 6 sets, and 1 minute rest between sets. Following the MWM application, Mulligan talus stabilization taping is performed. For this taping, the participants' ankles are placed on a stool at a height of 30 cm and their feet are placed in the dorsiflexion position. The therapist starts taping from the plantar surface of the calcaneus using rigid tape and will wrap and stabilize the talus.
  Arms: Intervention Group
Other: Sham — During joint mobilization with movement, the therapist will stabilize the ankle while performing knee flexion and ankle dorsiflexion by actively moving the center of mass to the affected side, but the shear force required to slide the tibia forward with the belt will not be given. Placebo taping following the application will be applied in such a way that there is no stabilization effect without tension between the same start and end points.
  Arms: Sham Group

SUMMARY:
Disorders caused by stroke may lead to significant limitations, especially in ankle range of motion, and may cause impairments in walking and balance functions. This limitation in ankle range of motion leads to difficulties in weight transfer, stability, and balance. As a result, there is a decrease in walking performance and an increased risk of falls. Various interventions have been used to improve ankle dorsiflexion passive range of motion, including gastrosoleus muscle stretching, muscle strengthening training, functional electrical stimulation training, proprioceptive control training, taping, manual therapy, different mobilization techniques, and ankle mobilization with motion (MWM).There are limited studies investigating the immediate effects of MWM and taping on gait and balance in stroke patients. This study was planned to investigate the effect of Mulligan's ankle MWM technique and talus stabilization taping on spatiotemporal gait and balance parameters in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

1. Having a unilateral stroke for more than three months,
2. Being able to walk 10 meters without an assistive device,
3. Being able to walk unassisted before having a stroke,
4. Having a score of 3 or lower on the Modified Ashworth Scale (MAS),
5. Be able to follow simple verbal instructions,
6. Being Volunteer

Exclusion Criteria:

1. Having had more than one stroke,
2. Cerebellar involvement,
3. Having severe visual impairment,
4. Having cognitive impairment,
5. Severe aphasia,
6. Apraxia,
7. Having contraindications for joint mobilization (e.g. ankle hypermobility, trauma, inflammation),
8. Have significant lower limb problems such as fractures or arthritis,
9. Having undergone musculoskeletal surgery less than 6 months ago,
10. Having joint contracture in the paretic ankle that prevents walking.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2024-02-14 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-10-11 (Actual)

PRIMARY OUTCOMES:
Stride length | Pre-intervention/sham and immediately after the intervention/sham
  Spatiotemporal parameters of gait will be evaluated with the Zebris FDM-2 device. Stride length spatiotemporal parameters of gait will be obtained from this platform. The date will recorded as a millimeter.
Stride width | Pre-intervention/sham and immediately after the intervention/sham
  Spatiotemporal parameters of gait will be evaluated with the Zebris FDM-2 device. Stride width spatiotemporal parameters of gait will be obtained from this platform. The date will recorded as a millimeter.
Cadance | Pre-intervention/sham and immediately after the intervention/sham
  Spatiotemporal parameters of gait will be evaluated with the Zebris FDM-2 device. Cadance spatiotemporal parameters of gait will be obtained from this platform. The date will recorded as the number of steps per minute.
Walking speed | Pre-intervention/sham and immediately after the intervention/sham
  Spatiotemporal parameters of gait will be evaluated with the Zebris FDM-2 device. Walking speed spatiotemporal parameters of gait will be obtained from this platform. The date will recorded as m/s.
The symmetry of the center of pressure changes during walking | Pre-intervention/sham and immediately after the intervention/sham
  Spatiotemporal parameters of gait will be evaluated with the Zebris FDM-2 device. The symmetry of the center of pressure changes during walking spatiotemporal parameters of gait will be obtained from this platform. The date will recorded as a millimeter.
The maximum force on the feet during walking | Pre-intervention/sham and immediately after the intervention/sham
  Spatiotemporal parameters of gait will be evaluated with the Zebris FDM-2 device. The maximum force on the feet during walking spatiotemporal parameters of gait will be obtained from this platform. The date will recorded as N/cm2.
The distribution of pressure on the feet | Pre-intervention/sham and immediately after the intervention/sham
  Spatiotemporal parameters of gait will be evaluated with the Zebris FDM-2 device. The distribution of pressure on the feet spatiotemporal parameters of gait will be obtained from this platform. The date will recorded as percentages.
Balance | Pre-intervention/sham and immediately after the intervention/sham
  Zebris FDM-2 device will also be used for the evaluation of balance parameters. Participants will be asked to stand on the device for 60 seconds without shoes, arms at their sides, eyes open and looking at a point 3 meters away. As a result of the evaluation, changes in the center of pressure will be recorded.

SECONDARY OUTCOMES:
10-meter walk test | Pre-intervention/sham and immediately after the intervention/sham
  The 10-meter walk test will be used to assess the walking speed of stroke patients. Patients will be asked to walk a 10-meter track. Walking times will be recorded in seconds.
Timed up and go test | Pre-intervention/sham and immediately after the intervention/sham
  The timed get up and walk test will be used to measure the dynamic balance of individuals. It includes the measurement of the time it takes for the participant to get up from the chair, walk 3 meters at their own pace, turn around, return to the chair and sit back in the chair.

CONTACTS AND LOCATIONS:
Overall Officials: İsmail Okur, Dr., Principal Investigator — Kutahya Health Sciences University
Locations (1):
- Kutahya Health Sciences University, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] An CM, Won JI. Effects of ankle joint mobilization with movement and weight-bearing exercise on knee strength, ankle range of motion, and gait velocity in patients with stroke: a pilot study. J Phys Ther Sci. 2016 Jan;28(2):689-94. doi: 10.1589/jpts.28.689. Epub 2016 Feb 29. PMID 27065565
- [Background] Altmis H, Oskay D, Elbasan B, Duzgun I, Tuna Z. Mobilization with movement and kinesio taping in knee arthritis-evaluation and outcomes. Int Orthop. 2018 Dec;42(12):2807-2815. doi: 10.1007/s00264-018-3938-3. Epub 2018 May 10. PMID 29750315
- [Background] An CM, Jo SO. Effects of Talocrural Mobilization with Movement on Ankle Strength, Mobility, and Weight-Bearing Ability in Hemiplegic Patients with Chronic Stroke: A Randomized Controlled Trial. J Stroke Cerebrovasc Dis. 2017 Jan;26(1):169-176. doi: 10.1016/j.jstrokecerebrovasdis.2016.09.005. Epub 2016 Oct 17. PMID 27765557